CLINICAL TRIAL: NCT04270721
Title: ESCP Safe Anastomosis proGramme in coLorectal surgEry
Acronym: EAGLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Birmingham (Other)
Collaborators: Ethicon, Inc. (Industry); European Society of Coloproctology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: RG_19196
Record Dates: First submitted 2019-12-12; First posted 2020-02-17 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Anastomotic Leak; Anastomosis; Complications
Keywords: anastomotic leak; right colectomy; cluster randomised study; leak prediction
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Intervention Model Description: EAGLE is an international, multicentre, cluster-sequence randomised controlled study. The intervention will be delivered at hospital-level so randomisation will be by hospital, with outcomes assessed at the individual patient level.
  Cluster randomisation will follow a dog-leg phased study design with 3 randomisation sequences. In the first phase, approximately 48 hospitals (clusters) are randomised between the three sequences, all three are eventually exposed to the intervention. Sequence 1 immediately receives the training intervention and data are only collected after the intervention. In sequence 2, data are collected before and after the intervention. The final sequence collects data only before the intervention. The second dogleg phase commences after the first when more clusters are ready to participate (indicatively after one month, but can be delayed as practicable). Indicatively, 7 dogleg phases with 48 hospitals each, will achieve the sample size required (333 clusters).
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient will be blinded to their hospital's randomised sequence allocation. Analysis will be performed blind to allocation sequence (and therefore before and after status) and after data have been cleaned and locked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- After intervention (sequence 1) (Experimental): 'After intervention' group receives the training immediately and data are only collected after the intervention.
  Interventions: Behavioral: The EAGLE Safe Anastomosis Quality Improvement Intervention
- Before and after intervention (sequence 2) (Experimental): For the 'Before and after intervention' group, data are collected both before and after the training.
  Interventions: Behavioral: The EAGLE Safe Anastomosis Quality Improvement Intervention
- Before intervention (sequence 3) (No Intervention): The 'before intervention' group collects data only before the training.
  *This arm will receive the educational intervention after data collection is completed.

INTERVENTIONS:
Behavioral: The EAGLE Safe Anastomosis Quality Improvement Intervention — The intervention is the same in each arm; the EAGLE Safe Anastomosis Quality Improvement Intervention is an educational programme for behavioural change composed of three parts:
  1. Introduction of a routine patient risk stratification for anastomotic leak
  2. Implementation of the ESCP Safe Anastomosis Checklist
  3. Adoption of a harmonised technique for stapled and handsewn anastomosis based on best evidence.
  Arms: After intervention (sequence 1); Before and after intervention (sequence 2)

SUMMARY:
EAGLE is an international service improvement study to investigate the value of an educational tool delivered to surgeons and their teams to reduce the risk of anastomotic leak (leak of a join in the bowel) after right hemicolectomy or ileocaecal resection. This complication causes significant risk to life and therefore risks of leak should be minimised.

The educational team of the European Society of Coloproctology has developed an online training package to deliver to 350 hospitals in 30 countries.

DETAILED DESCRIPTION:
EAGLE is an international quality improvement programme to share best practice and harmonise ileo-colic anastomosis procedures through an education programme for surgeons and theatre teams.

The programme has 3 main strategies: (i) enhanced pre-operative risk stratification (making sure it is safe to join the bowel together for each patient); (ii) harmonisation of surgical technique (making the join as good as it can be and checking it carefully after it is created), and (iii) implementation of an intra-operative anastomosis 'checklist' (focusing the attention of the whole theatre team at this critical stage of the operation). The investigators will use a novel scientific approach to assess the patient benefit that enables not only the quality improvement itself to be delivered to all participating hospitals but also enables collection and analysis of data to measure the effect of these measures. The best way of doing this is to embed the proposed quality improvement into a staggered implementation programme, allowing the effect to be assessed between the centres. The specific methodology proposed introduces the intervention in a step-wise fashion to all hospitals. By the end, all sites will have implemented the programme. Overall, the investigators hope to reduce the leak rate by 30% from 8.1% to 5.6% in about 4,500 patients.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (age 18 years and above) undergoing right colectomy with or without primary anastomosis. Right colectomy is defined as ileocaecal resection or right hemicolectomy (any colonic transection with the distal resection margin proximal to the splenic flexure).
* All patients undergoing right colectomy are eligible, including those who do not have an anastomosis and are defunctioned by a proximal stoma.
* Procedures for any pathology, via any operative approach (open, laparoscopic, robotic or converted) are eligible.
* Elective (surgery on a planned admission), expedited, and emergency (surgery on an unplanned admission) procedures are eligible.

Exclusion Criteria:

* Patients undergoing more than one gastrointestinal anastomosis during the same operation.
* In Crohn's disease, additional upstream stricturoplasty or resection/anastomosis to treat disease or strictures at the same operation.
* Simultaneous right colectomy and hyperthermic intraperitoneal chemotherapy (HIPEC) and/or cytoreductive surgery.
* Each individual patient should only be included in EAGLE once. Following the index procedure that is included in EAGLE, patients undergoing additional procedures within the study window should not be included for a second time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4400 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients diagnosed clinically or radiologically with anastomotic leak within 30 days of surgery | up to 30 days from operation
  Anastomotic leak is defined as anastomotic leak identified radiologically or clinically, or intra-peritoneal (abdominal or pelvic) fluid collection identified radiologically, as per the Centre for Disease Control Criteria for Organ Space infection.
  This will be described as a rate divided by the total number of patients who had a primary anastomosis (rather than total number of patients undergoing right hemicolectomy or ileocaecal resection).

SECONDARY OUTCOMES:
The rate of re-operation for anastomotic leak | up to 30 days
  The number of patients re-operated, of those diagnosed with anastomotic leak following right hemicolectomy or ileocaecal resection
The rate of adverse outcomes following right hemicolectomy or ileocaecal resection | up to 30 days
  For all patients included in the study (i.e. who underwent right hemicolectomy or ileocaecal resection whether or not with primary anastomosis);
  1. Number of patients undergoing re-operation for any cause within 30 days
  2. Number of patients with unplanned admission to critical care within 30 days
  3. Number of patients re-admitted to hospital within 30 days
  4. Mortality rate within 30 days
The rate of stoma formation | At index operation
  For all patients included in the study (i.e. who underwent right hemicolectomy or ileocaecal resection whether or not with primary anastomosis);
  1. Rate of formation of ileostomy without primary anastomosis
  2. Rate of defunctioning ileostomy with primary anastomosis
Length of hospital stay following right hemicolectomy or ileocaecal resection | up to 30 days
  Measured in post-operative days

OTHER OUTCOMES:
Feasibility of recruitment of clusters (hospitals) in this study design | Through to study completion, expected 1 year
  Measured by the number of participating hospitals and countries
Time to site set-up in this study design | Through to study completion, expected 1 year
  Time taken for study set-up at sites from registration to randomisation
Uptake of online educational modules | Through to study completion, expected 1 year
  The proportion of eligible surgeons to undertake the educational modules in participating units.
Understanding uptake and effectiveness of online educational modules | Surgeons will have 30 days to complete the educational evaluation to collect CPD (continuing professional development) certificate. Interviews will take place 3-6 months after study completion at individual units.
  Semi-structured interviews will be undertaken at purposefully sampled units to assess longevity of the intervention
Adherence to implementation of the Safe Anastomosis Programme | day of index operation
  The proportion of eligible patients whose team completed the pre-operative risk stratification and Safe Anastomosis Checklist

CONTACTS AND LOCATIONS:
Overall Officials: Dion Morton, Principal Investigator — University of Birmingham
Locations (1):
- Clinic of Coloproctology and Minimally Invasive Surgery, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
The investigators anticipate that the study protocol will be published early 2020. The Clinical Study report will be published most likely in 2021.
  This study will not collect patient identifiable data. All 'individual participant data' will be anonymised.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available beginning 6 months and ending 36 months after the primary study analysis has been published.
Access Criteria: Data will be available to researchers submitting a methodologically sound proposal. Proposals should be directed to Dion.Morton@uhb.nhs.uk. To gain access requestors will need to sign a data access agreement.
  After 36 months the data will be available but without investigator support other than deposited metadata.

REFERENCES:
- [Derived] ESCP EAGLE Safe Anastomosis Collaborative and NIHR Global Health Research Unit in Surgery. Evaluation of a quality improvement intervention to reduce anastomotic leak following right colectomy (EAGLE): pragmatic, batched stepped-wedge, cluster-randomized trial in 64 countries. Br J Surg. 2024 Jan 3;111(1):znad370. doi: 10.1093/bjs/znad370. PMID 38029386
- [Derived] Venn ML, Knowles CH, Li E, Glasbey J, Morton DG, Hooper R; ESCP EAGLE Safe Anastomosis Collaborative. Implementation of a batched stepped wedge trial evaluating a quality improvement intervention for surgical teams to reduce anastomotic leak after right colectomy. Trials. 2023 May 15;24(1):329. doi: 10.1186/s13063-023-07318-9. PMID 37189166
- [Derived] ESCP EAGLE Safe Anastomosis Collaborative. ESCP Safe Anastomosis ProGramme in CoLorectal SurgEry (EAGLE): Study protocol for an international cluster randomised trial of a quality improvement intervention to reduce anastomotic leak following right colectomy. Colorectal Dis. 2021 Oct;23(10):2761-2771. doi: 10.1111/codi.15806. Epub 2021 Aug 25. PMID 34255417